CLINICAL TRIAL: NCT01051388
Title: Prophylactic Efficacy of Proton Pump Inhibitor on Recurrence of Peptic Ulcer in Patients Continuously Treated With Low-dose Aspirin-Randomized, Multi-center, Single-blinded, Parallel-group, Comparative Study
Brief Title: Cardio-cerebrovascular Disease and Aspirin Ulcer Relapse Evaluation
Acronym: CARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Gastro-Intestinal Medical Care Research Center (Unknown)
Responsible Party: Takeshi Azuma, Kobe University, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TRIGID0801; UMIN000002901 (Other: Japan: Infrastructure for Academic Activities, University hospital Medical Information Network)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Cardio-cerebrovascular Disease
Keywords: The efficacy of PPI; Patients receiving low-dose aspirin for vascular protection
MeSH Terms: interventions — Rabeprazole; Gefarnate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Active Comparator): Low-dose PPI (Rabeprazole sodium 10 mg)
  Interventions: Drug: Low-dose PPI (Rabeprazole sodium)
- Group II (Active Comparator): High-dose PPI (Rabeprazole sodium 20 mg)
  Interventions: Drug: High-dose PPI (Rabeprazole sodium)
- Group III (Active Comparator): Non-PPI (Gefarnate)
  Interventions: Drug: Non-PPI (Gefarnate)

INTERVENTIONS:
Drug: Low-dose PPI (Rabeprazole sodium) — PPI (Rabeprazole sodium 10 mg), once a day, for four weeks times three
  Arms: Group I
Drug: High-dose PPI (Rabeprazole sodium) — PPI (Rabeprazole sodium 20 mg Tablet once a day, for four weeks times three)
  Arms: Group II
Drug: Non-PPI (Gefarnate) — The mucosal defensive drug (Gefarnate 50 mg Capsule, twice a day, for four weeks times three)
  Arms: Group III

SUMMARY:
The aim of this study is to evaluate the efficacy of proton pump inhibitor (PPI), comparing to the mucosal defensive drug, in the prevention of the recurrence of gastric and/or duodenal ulcers during 12 weeks observation in patients receiving low-dose aspirin for vascular protection.

DETAILED DESCRIPTION:
The events of recurrence of gastric and/or duodenal ulcers will be evaluated due to a blinded manner by specialized endoscopists at pre- and post administration during 12 weeks administration of PPI (Rabeprazole sodium 10 mg or 20 mg tablet once a day) or the mucosal defensive drug (Gefarnate 50mg Capsule twice a day).

ELIGIBILITY:
Inclusion Criteria:

* patients with ischemic heart failure or vascular disease of brain
* patients taking low-dose aspirin to prevent relapse of vascular diseases
* patients who experienced gastric and/or duodenal ulcers before the study by the endoscopy
* patients without active gastric and duodenal ulcers
* more than 20 years old
* outpatients
* patients written an informed consent

Exclusion Criteria:

* patients with ischemic heart failure, which are acute phase, unstable condition or under 6 months after stent-instillation
* patients with brain vascular disease , which are acute phase, unstable condition or under 3 months after the first attack
* patients who are uncontrolled and complicated disease, for example thrombocytopenia, and unsuitable for this study as judged by investigator
* patients who are treated with steroid hormones
* patients who are women of, pregnant and lactating and childbearing
* patients who are alcoholism
* patients who show the hypersensitivity for test drugs
* patients who are enrolled in another clinical study
* patients who are judged as unsuitable by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Endoscopic Recurrence of Gastric and/or Duodenal Ulcers | 12 weeks after giving medication

SECONDARY OUTCOMES:
Recurrence of gastrointestinal mucosal lesions, Lanza score and its changes form baseline, and incidences of adverse events | 12 weeks after giving medication

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Azuma, M.D., Ph.D., Principal Investigator — Kobe University, School of Medicine
Locations (1):
- Kobe University, School of Medicine, Kobe, Hyōgo, Japan

REFERENCES:
- See also: Related Info — https://upload.umin.ac.jp/cgi-open-bin/ctr/ctr.cgi?function=brows&action=brows&type=summary&recptno=R000003537&language=J